CLINICAL TRIAL: NCT06274957
Title: The Effect of Airway Oscillation and Chest Wall Oscillation on Respiratory Functions and Sleep Quality in COPD Patients in Acute Exacerbation Period and Technical Inspection of Devices
Brief Title: The Effect of Airway and Chest Wall Oscillation on Respiratory Functions in COPD Patients in Acute Exacerbation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gamze Altınkaynak, Principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SaglikBilimleriUN
Record Dates: First submitted 2024-02-02; First posted 2024-02-23 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: COPD Exacerbation Acute
Keywords: copd; pep; hfcwo; airway clearance techniques
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Experimental): Conventional training was applied to the patients
  Interventions: Other: CONTROL
- Positive Expiratory Pressure (Experimental): We applied PEP (positive expiratory pressure) therapy in adddition to the conventional exercises
  Interventions: Device: PEP DEVICE
- High Frequency Chest Wall Oscillation (Experimental): We applied HFCWO (High Frequency Chest Wall Oscillation) in addition to the conventional exercises
  Interventions: Device: HFCWO DEVICE

INTERVENTIONS:
Other: CONTROL — Pursed Lips breathing exercise, Active Respiratory Techniques Cycle, Postural Drainage, Mobilization, Calisthenic Exercises, and Patient Education. Relaxation positions and energy conservation techniques were taught in Patient Education
  Arms: control
Device: PEP DEVICE — Pursed Lips breathing exercise, Active Respiratory Techniques Cycle, Postural Drainage, Mobilization, Calisthenic Exercises, and Patient Education. Relaxation positions and energy conservation techniques were taught in Patient Education
  PEP training was applied using the Acapella device.
  In addition, participants were subjected to two sessions of 10 minutes each with the Acapella device. In the study, the Acapella device, capable of sustaining expiratory flow of at least 15 L/min for 3 seconds, was activated by taking a deep breath, holding the breath for 2-3 seconds, and then exhaling into the device.
  Arms: Positive Expiratory Pressure
Device: HFCWO DEVICE — Patients were provided with conventional exercises including Pursed Lips breathing exercise, Active Respiratory Techniques Cycle, Postural Drainage, Mobilization, Calisthenic Exercises, and Patient Education. Relaxation positions and energy conservation techniques were taught in Patient Education
  In addition, participants will receive High-Frequency Chest Wall Oscillation (HFCWO) therapy twice a day for 10 minutes each.
  HFCWO training was applıed using the WEST device
  Arms: High Frequency Chest Wall Oscillation

SUMMARY:
Chronic obstructive pulmonary disease (COPD); It is a common, treatable and preventable disease characterized by progressive and irreversible airflow limitation and has systemic effects with respiratory system involvement. Increased respiratory workload, decreased work .

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD); It is a common, treatable and preventable disease characterized by progressive and irreversible airflow limitation and has systemic effects with respiratory system involvement. Increased respiratory workload, decreased work of breathing in patients are important factors that cause respiratory and peripheral muscle strength and functional capacity exercise intolerance. It is defined as an exacerbation if there is an increase in shortness of breath, cough, sputum amount and purulence, which necessitates a change in treatment in the COPD patients. In the guides; Individualized exercise training for disease management is an essential component of these programs. In the literature; Although there are many studies showing the beneficial effects of traditional exercise training programs in patients with COPD, physiotherapy applications used in the exacerbation period are recommended, but there are not many studies examining the device technologies used in this area. In this period, devices that provide chest wall oscillation and airway oscillation can be preferred for the symptomatic treatment of increasing cough and sputum complaints. There is no study comparing these two methods that we know of. Our study will be carried out on 33 patients hospitalized in the Pulmonology Service of the Health Sciences University Gülhane Training and Research Hospital, followed up with the diagnosis of COPD exacerbation, who met the inclusion criteria and accepted to participate in the study on a voluntary basis. Patients will be randomized into 3 groups as 2 experiments and 1 control. Measurements of patients admitted to the ward will be made at the beginning and end of the study. Socio-demographic data of the patient, chest circumference measurement, COPD assessment test, mMRC dyspnea scale, BODE index, pulmonary function test, arterial blood gas, chest X-ray, 30-second sit and stand test, Richard-Campbell Sleep Scale, Clinical COPD Questionnaire, Charlson comorbidity index will be applied. Pursed-lip breathing, active breathing techniques cycle, bronchial hygiene techniques, mobilization, calisthenic exercises and patient education (teaching relaxation positions and energy conservation techniques) will be applied to the patients in the study and control groups during their hospitalization. Chest wall oscillation will be practiced together with chest physiotherapy in the 1st experimental group, and airway oscillation will be practiced in the 2nd experimental group with the same physiotherapy program. In the study, the clinical use and technical features of the devices will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Being classified as GOLD stage 3 or 4 based on spirometric evaluation in the medical history.
* Having a hospital admission within the specified time frame, evaluated by a pulmonary specialist, and admitted to the pulmonary diseases service with a diagnosis of COPD exacerbation.
* Being 40 years of age or older.
* Voluntarily agreeing to participate in the study.

Exclusion Criteria:

* Having a hospital admission with a diagnosis of asthma attack in the last 5 years.
* Monitoring suspicious focal points for pneumonia on lung radiology.
* Hospitalization due to reasons other than exacerbation despite having a diagnosis of COPD.
* Presence of pulmonary fibrosis or suspicious findings of fibrosis on radiology.
* Systemic fungal infections.
* Having cognitive impairment affecting the decision to participate in the study, such as confusion, orientation disorder, or dementia.
* Patients with lung cancer or metastasis in the lungs.
* Diagnosis of conditions provoking shortness of breath other than COPD exacerbation, such as pneumonia, pneumothorax, heart failure, and pulmonary embolism.
* Presence of a new-onset rhythm disorder or ischemic changes requiring intervention on the EKG, excluding sinus tachycardia and multifocal atrial tachycardia.
* Chronic kidney failure requiring hemodialysis.
* Patients with conditions causing weakness in the lower extremities, such as arthritis, neurological disease, deep vein thrombosis, peripheral artery disease, muscle weakness, fractures, osteoarthritis, etc.
* Having ankylosing spondylitis with a Cobb angle of 10 degrees or more in the radiographic evaluation of the vertebral column.
* Having undergone surgery on the upper extremities, lower extremities, neck, and back.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-17 (Estimated)

PRIMARY OUTCOMES:
COPD assessment test | The first and last day of the training will be measured an avarage 7 days
  The COPD assessment test (CAT) includes eight items related to the severity of dyspnea, exercise capacity, cough, sputum, chest tightness, sleep quality, self-confidence, and energy levels. The CAT is a short and simple instrument to evaluate COPD patients, and its validated translations are present in a broad range of languages in the world. Additionally, the CAT is correlated with quality of life. According to the GOLD guidelines, patients with CAT score of ≥10 or mMRC score of ≥2 represents have more prominent symptoms. The cutoff points of more symptoms for CAT score ≥10 was validated in COPD. This threshold has been detected to have an important impact on the daily lives of patients with COPD.
Clinical COPD Questionnaire | The first and last day of the training will be measured an avarage 7 days
  The Clinical COPD Questionnaire, developed by Thys Van der Molen, consisting of 10 items (4 items for symptoms, 4 items for functional status, and 2 items for mental status) assessing clinical control for the purpose of evaluating functional status, mental status, and symptoms, will be administered to all cases. In a study conducted by Reda and colleagues in 2010, it was demonstrated that the Clinical COPD Questionnaire is a valid, reliable, and sensitive tool for use in individuals at risk of COPD and in COPD patients
mMRC dyspnea scale | The first and last day of the training will be measured an avarage 7 days
  The perception of dyspnea in patients will be assessed using the mMRC dyspnea scale. This scale, modified by ATS, evaluates dyspnea and limitations in daily life activities. Patients are asked to choose the most suitable expression from the five statements ranging from '0-4' (0: Only shortness of breath during heavy exercise; 4: Being housebound due to breathlessness, experiencing shortness of breath even during light activities such as dressing and undressing) to describe their own perception of dyspnea. The scale developed by Richards in 1987 consists of 6 items assessing the depth of nocturnal sleep, sleep onset latency, frequency of awakening, duration of wakefulness upon awakening, sleep quality, and ambient noise level. Each item is evaluated on a visual analog scale ranging from 0 to 100. Scores between "0-25" indicate very poor sleep, while scores between "76-100" indicate very good sleep. The scale's total score is assessed based on 5 items, excluding the 6th item evaluating
Richard-Campbell Sleep Questionnaire | The first and last day of the training will be measured an avarage 7 days
  The scale developed by Richards in 1987 consists of 6 items assessing the depth of nocturnal sleep, sleep onset latency, frequency of awakening, duration of wakefulness upon awakening, sleep quality, and ambient noise level. Each item is evaluated on a visual analog scale ranging from 0 to 100. Scores between "0-25" indicate very poor sleep, while scores between "76-100" indicate very good sleep. The scale's total score is assessed based on 5 items, excluding the 6th item evaluating ambient noise level from the overall score. As the score on the scale increases, patients' sleep quality also improves. The Cronbach's alpha value for the scale, developed by Richards, was found to be 0.82. The Turkish validity and reliability of the scale were conducted by Özlü and Özer, revealing a Cronbach's alpha value of 0.91
30 second sit and stand | The first and last day of the training will be measured an avarage 7 days
  test is primarily used for evaluating function and physical performance associated with mobility, and is suggested as an acceptable alternative method for assessing functional capacity in COPD. The patient, who has received medical treatment in an environment equipped with a chair with a seat height of approximately 44 cm and a backrest, preferably without armrests, a stopwatch, oxygen support if needed, a blood pressure monitor, and a defibrillator, and has not engaged in heavy activity in the last 2 hours, will be explained the test procedure in a comprehensible manner. Resting blood pressure, oxygen saturation, pulse, and modified Borg dyspnea score will be recorded. The patient will be instructed to cross their arms and touch both shoulders, then sit and stand up from the chair for 30 seconds in this position. At the end of the test, blood pressure, oxygen saturation, pulse, modified Borg dyspnea score, and the number of sit-to-stand repetitions within 30 seconds will be record
BODE index | The first and last day of the training will be measured an avarage 7 days
  The BODE index has been developed to assess the mortality risk in patients with COPD. The BODE index comprises parameters such as BMI (Body Mass Index), the severity of airflow limitation, perceived degree of dyspnea, and exercise capacity. BMI will be calculated using the weight/height² formula, the severity of airflow limitation will be assessed by FEV1 % predicted, the perceived degree of dyspnea will be evaluated using the mMRC scale, and exercise capacity will be determined with the 6MWT (6-Minute Walk Test) in patients with COPD.
chest circumference measurements | The first and last day of the training will be measured an avarage 7 days
  To assess chest mobility and respiratory type, chest circumference measurements will be taken using a tape measure at axillary (at the level of the 4th rib), epigastric (at the xiphoid process level), and subcostal (above the 11th and 12th ribs) regions. Measurements will be taken in an upright sitting position, during neutral, deep inspiration, and deep expiration. The difference between deep inspiration and deep expiration will be recorded in centimeters
Modified Borg Scale | The first and last day of the training will be measured an avarage 7 days
  This scale was developed by Borg in 1970 for the purpose of measuring the perceived exertion during physical exercise. It is commonly used to assess the intensity of dyspnea during effort and at rest. Comprising ten grades that describe the severity of dyspnea, the Modified Borg Scale (MBS) makes it easier for patients by providing clear definitions for the intensity of dyspnea
muscle strenght test | The first and last day of the training will be measured an avarage 7 days
  Muscle strength testing is used to determine the capability of the muscle or muscle group to produce force. It provides information that is useful in differential diagnosis, prognosis and management of neuromuscular and musculoskeletal disorders. its evaluating muscle strength is the Oxford Scale (AKA Medical Research Council Manual Muscle Testing scale). This method involves testing key muscles from the upper and lower extremities against the examiner's resistance and grading the patient's strength on a 0 to 5 scale accordingly

CONTACTS AND LOCATIONS:
Overall Officials: ZUHAL KUNDURACILAR, PROF. DR., Study Director — SAGLIK BILIMLERI UNI; GAMZE KOYUTURK, PT, PHD (C), Principal Investigator — SAGLIK BILIMLERI UNI; AYSUNA DINCER, DOCTOR, Study Chair — SAGLIK BILIMLERI UNI; MEHMET YUKSEKKAYA, ASIST PROF, Study Chair — ANKARA UNI
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)